CLINICAL TRIAL: NCT02974192
Title: Neoptrin, Soluble CD40-ligand and Ischemic Stroke: a Clinical Perspective
Brief Title: Neopterin Effects on Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate profossor of anesthesia, Assiut University
Other Study IDs: IIRB0000871432
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Stroke
Keywords: Ischemic stroke; Soluble CD40 Ligand; Neopetrin; stroke risk factors; functional outcome
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Neopterin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Neopterin — Neopterin will be measured by using standard laboratory methods on the first day of admission.

SUMMARY:
Ischemic stroke accounts for the majority of stroke cases and constitutes a major cause of death and disability in industrial world. Inflammation has been reported to constitute a major component of ischemic stroke pathology. The brain responds to ischemic injury with an acute andprolonged inflammatory process. Few studies have investigated the relationship between acute biomarkers of inflammation and functional outcome following stroke

DETAILED DESCRIPTION:
This case -control observational prospective study will be conducted on 100 patients with first -ever acute onset ischemic stroke within 24-48 hours. Their ages ranged-years old (mean age ±years). All participants will be subjected to thorough history taking, full clinical and neurological examination. Complete neurological examination where the following clinical and demographical data will be taken; age sex, stroke etiology, presence of stroke risk factors (as smoking history , hyperlipidemia, diabetes mellitus , history of hypertension, history of transient ischemic attacks, history of myocardial infarction or any cardiac problems). Stroke subtype will be classified according to the criteria of Trial of Org 10172 in acute Stroke Treatment (TOAST) classification. The clinical stroke syndrome will be determined by applying the criteria of the Oxfordshire Community Stroke project (OCSP). Stroke severity will be assessed by Scandinavian Stroke Scale (SSS) and Modified Rankin Scale (mRS) will be measured at the time of admission. Brain imaging (either CT scan and /or MRI) will be performed after admission. Electrocardiography (ECG), Echocardiography (ECHO), Carotid and vertibrobasilar Duplex will be done for all patients. Blood samples will be drawn for assessment of complete blood picture (CBC), Random blood glucose levels, renal function tests (RFT), liver function tests (LFT), thyroid function tests (TFT), Lipid profile, Soluble CD40 Ligand and Neopetrin by using standard laboratory methods on the first day of admission.

ELIGIBILITY:
Inclusion Criteria:

* Onset is within one week
* Confirmed stroke by brain CAT and / or MRI scan infarction
* Exclusion Criteria:
* Cognitive and mental changes
* Recurrent stroke
* Hepatic and renal impairment
* Endocrinal diseases
* Steroid therapy
* Previous fractures
* brain neoplasm,
* Autoimmune diseases
* History of acute and chronic inflammatory diseases
* Malignancy,
* Trauma
* Surgery
* Acute vascular diseases that occurred within four weeks prior the onset of stroke History myocardial infarction ˂3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with first -ever acute onset ischemic stroke within 24-48 hours
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Neopterin level | Within the first 24 hours
  will be measured by using standard laboratory methods on the first day of admission
Soluble CD40 Ligand | Within the first 24 hours
  will be measured by using standard laboratory methods on the first day of admission

SECONDARY OUTCOMES:
Stroke subtype | Within the first 24 hours
  will be classified according to the criteria of Trial of Org 10172 in acute Stroke Treatment (TOAST) classification
The clinical stroke syndrome | Within the first 24 hours
  will be determined by applying the criteria of the Oxfordshire Community Stroke project (OCSP)
Stroke severity | Within the first 24 hours
  Stroke severity will be assessed by Scandinavian Stroke Scale (SSS) and Modified Rankin Scale (mRS) will be measured at the time of admission.

CONTACTS AND LOCATIONS:
Overall Officials: Sayed k Abd-Elshafy, MD, Principal Investigator — Associate professor of anesthesia
Locations (1):
- Faculty of Medicine, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided